CLINICAL TRIAL: NCT01140022
Title: Leveraging Technology as a Clinician Extender to Screen Culturally Diverse Young Women for Chlamydia
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H1095-31344
Record Dates: First submitted 2010-05-18; First posted 2010-06-09 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Chlamydia; Screening
Keywords: Chlamydia, Screening, young women, kiosk, computer module
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female Patients 18-25 yo: Female patients aged 18-25 who have come to one of the ED or urgent care sites for care, regardless of the presence of CT symptoms.
  Interventions: Other: CT Screening

INTERVENTIONS:
Other: CT Screening — Patients will use a kiosk module that will provide information about CT screening and assess their risk for CT. Patients choosing to get a CT screening will receive a printout instructing the provider or nurse to collect a urine sample for CT screening.

SUMMARY:
The purpose of this study is to conduct a quality improvement intervention to improve the ability of health care providers to deliver an important preventive health service (CT screening) in order to meet the goal of universal CT screening for young women age 25 or younger as recommended by the CDC and virtually all major health organizations. This novel approach utilizes a bilingual (English-Spanish) computer kiosk module to deliver education about CT and allow patients to request a CT screening test. This module should significantly increase CT screening among at risk women (18-25yo) attending urgent care clinics and emergency departments.

DETAILED DESCRIPTION:
Chlamydia trachomatis (CT) remains epidemic among sexually young adult and adolescent females especially ethnic minority women. Despite recommendations for at least annual screening of all sexually active women up to age 25, CT screening rates remain low. Most young women do not regularly attend primary care clinics where preventive care such as CT screening should be done; and clinicians lack time and comfort to address CT screening during the context of an urgent care or emergency department visit. This proposed study takes advantage of a "missed opportunity" for screening these at-risk young women for CT when they come in contact with the health care system during an urgent care or emergency department visit. The purpose of this study is to conduct a quality improvement intervention, to improve the ability of health care providers to deliver an important preventive health service (CT screening) in order to meet the goal of universal CT screening recommended by virtually all major health organizations. CT screening should be done as a routine part of health care but currently is not. In this study, we will help providers do what they should already be doing using this novel health care delivery approach. In this study, we created and are evaluating a bilingual (English-Spanish) computer kiosk module to increase CT screening among at risk English and Spanish speaking women (18-25 yo) attending urgent care clinics and emergency departments (ED). This computer technology will be able to conduct many of the steps necessary for CT screening including assessing clients' CT risk and prompting the client and health care professionals for CT urine specimen collection. This study will also examine the extent to which this computer kiosk module intervention use is acceptable and feasible among both English and Spanish speaking young women, and health care professionals who care for them in urgent care and ED settings. This type of intervention to improve CT screening is potentially translatable to a wide variety of health delivery settings as it is not dependent on staff time, motivation or skill to assess sexual history in the busy urgent care setting. This project also supports current recommendations of Healthy People 2010, the U.S. Preventive Services Task Force and other professional organizations to screen all sexually active young adult females at least annually for CT to address this important public health problem especially among our young ethnic minority women who carry the largest STI disease burden. Early detection through routine CT screening coupled with appropriate treatment of CT infections can eliminate widespread infection and prevent such major reproductive morbidity.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Medically Stable
* Sexually active
* Female
* 18-25 years old
* Seeking health services in participating urgent care clinics and ED in San Francisco/Bay Area, California.

Exclusion Criteria:

* Clients who do not speak English or Spanish will not be eligible to participate.
* Males of any age because there is no CDC recommendation to universally screen this group.
* Women who have never had sexual intercourse are not eligible as this is a study of how to increase screening for chlamydia, a sexually transmitted infection.
* For Kiosk, clients with moderate and major trauma or illness requiring immediate medical intervention, as assessed by triage nurse as part of routine protocol, will be excluded from participation.
* Anyone who chooses not to participate (as this is voluntary) will be excluded from participation.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients 18-25 yo receiving care at urgent care or ED sites.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proportion of female patients 18-25yo receiving CT screening during ED or UC visit. | one year prior to the patient's clinic or ED visit.

SECONDARY OUTCOMES:
Acceptability of module and intervention among patients and staff. | one year prior to the patient's clinic or ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ann Shafer, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - CMC Fresno Emergency Department, Fresno, California
  - Alameda County Medical Center, Highland Hospital, Oakland, California
  - San Francisco General Hospital - Emergency Department, San Francisco, California
  - San Francisco General Hospital, Urgent Care, San Francisco, California
  - UCSF Emergency Deparmtent, San Francisco, California
  - UCSF Screening and Acute Care Clinic, San Francisco, California